CLINICAL TRIAL: NCT05158751
Title: Myocarditis Causing Premature Ventricular Contractions:Insights From the MAVERIC Registry
Acronym: MAVERIC
Status: Not yet recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRF-MAVERIC REG-0009
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-10

CONDITIONS: Myocarditis; Premature Ventricular Contractions; Ventricular Tachycardia (VT)
MeSH Terms: conditions — Myocarditis; Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess potential link between unrecognized myocardial inflammation (myocarditis) and premature ventricular contractions (PVCs) associated with and without reduced Left ventricular ejection fraction (LVEF) through comprehensive diagnostic work up.

DETAILED DESCRIPTION:
Hypothesized that occult inflammation is clinically under-recognized in patients with symptomatic PVCs with and without Left ventricular (LV) dysfunction and can be a potential link between the 2 conditions. Aimed to evaluate the incidence of underlying inflammation using the Positron emission tomography (PET) scan in patients presenting with symptomatic PVCs enrolled retrospectively in the MAVERIC registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age with mono-morphic or polymorphic PVC burden of ≥5000 in 24 hours.
* Non-sustained VT was defined as ≥3 more consecutive beats lasting <30 seconds

Exclusion Criteria:

* History of myocardial infarction,
* Significant flow-limiting coronary artery disease (≥50% stenosis) on invasive coronary angiography or CT angiography,
* History of revascularization,
* Significant symptomatic atrial arrhythmias associated with LV dysfunction,
* Severe valvular disease,
* Cardiomyopathy attributed to toxins such as alcohol and illicit drugs,
* History of cardiac arrest,
* History of channelopathies or inherited arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females with PVC and ventricular tachycardia (VT) will be enrolled if they meet the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Identify the underlying myocarditis in patients presenting with PVCs with or without reduced LVEF | Retrospective Collection between dates January 2014-January 2023
  To identify the underlying myocarditis in patients presenting with PVCs with or without reduced LVEF through laboratory testing, FDG-PET(18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose - positron emission tomography) scan, Cardiac Magnetic Resonance imaging and/or Endomyocardial biopsy.

SECONDARY OUTCOMES:
Ascertain whether immunosuppressive therapy (IST) affords short term and long term improvement of LVEF and clinical outcomes | Retrospective Collection between dates January 2014-January 2023
  To ascertain whether immunosuppressive therapy (IST) affords short term and long term improvement of LVEF and clinical outcomes in virus negative and FDG-PET positive patients with non-ischemic cardiomyopathy, myocardial inflammation and PVCs.

OTHER OUTCOMES:
Evaluate whether IST + catheter ablation results in optimal clinical response | Retrospective Collection between dates January 2014-January 2023
  To evaluate whether IST + catheter ablation results in optimal clinical response in virus negative and FDG-PET positive patients with PVCs with or without reduced LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

REFERENCES:
- [Background] Ahn MS. Current Concepts of Premature Ventricular Contractions. J Lifestyle Med. 2013 Mar;3(1):26-33. Epub 2013 Mar 31. PMID 26064834
- [Background] Ng GA. Treating patients with ventricular ectopic beats. Heart. 2006 Nov;92(11):1707-12. doi: 10.1136/hrt.2005.067843. No abstract available. PMID 17041126
- [Background] Kennedy HL, Whitlock JA, Sprague MK, Kennedy LJ, Buckingham TA, Goldberg RJ. Long-term follow-up of asymptomatic healthy subjects with frequent and complex ventricular ectopy. N Engl J Med. 1985 Jan 24;312(4):193-7. doi: 10.1056/NEJM198501243120401. PMID 2578212
- [Background] Lakkireddy D, Turagam MK, Yarlagadda B, Dar T, Hamblin M, Krause M, Parikh V, Bommana S, Atkins D, Di Biase L, Mohanty S, Rosamond T, Carroll H, Nydegger C, Wetzel L, Gopinathannair R, Natale A. Myocarditis Causing Premature Ventricular Contractions: Insights From the MAVERIC Registry. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007520. doi: 10.1161/CIRCEP.119.007520. Epub 2019 Dec 16. PMID 31838913
- [Background] Ruberman W, Weinblatt E, Goldberg JD, Frank CW, Shapiro S. Ventricular premature beats and mortality after myocardial infarction. N Engl J Med. 1977 Oct 6;297(14):750-7. doi: 10.1056/NEJM197710062971404. PMID 70750
- [Background] Whiting RB. Ventricular premature contractions. Which should be treated? Arch Intern Med. 1980 Nov;140(11):1423-6. PMID 6159832
- [Background] Piccolo E, Raviele A. [Clinical and prognostic significance of hyperkinetic ventricular arrhythmias]. G Ital Cardiol. 1983;13(4):276-89. Italian. PMID 6350092
- [Background] Kastor JA. Ventricular premature beats. Adv Intern Med. 1983;28:63-91. PMID 6340432
- [Background] Wu AH. Management of patients with non-ischaemic cardiomyopathy. Heart. 2007 Mar;93(3):403-8. doi: 10.1136/hrt.2005.085761. No abstract available. PMID 17322525
- [Background] Tschope C, Cooper LT, Torre-Amione G, Van Linthout S. Management of Myocarditis-Related Cardiomyopathy in Adults. Circ Res. 2019 May 24;124(11):1568-1583. doi: 10.1161/CIRCRESAHA.118.313578. PMID 31120823
- [Background] Mattsson G, Magnusson P. Electrical storm in the inflamed heart: ventricular tachycardia due to myocarditis. Clin Case Rep. 2017 Jul 3;5(8):1327-1332. doi: 10.1002/ccr3.1071. eCollection 2017 Aug. PMID 28781852
- [Background] Ms Alina Scridon Mr Philippe Chevalier , FESC. Ventricular arrhythmias complicating acute myocarditis. ESC Council for Cardiology Practice Vol. 9, N° 26 - 05 Apr 2011
- [Background] Frustaci A, Priori SG, Pieroni M, Chimenti C, Napolitano C, Rivolta I, Sanna T, Bellocci F, Russo MA. Cardiac histological substrate in patients with clinical phenotype of Brugada syndrome. Circulation. 2005 Dec 13;112(24):3680-7. doi: 10.1161/CIRCULATIONAHA.105.520999. PMID 16344400
- [Background] Salerno F, Girerd N, Chalabreysse L, Billaud G, Lina B, Chevalier P. Myocarditis and cardiac channelopathies: a deadly association? Int J Cardiol. 2011 Mar 17;147(3):468-70. doi: 10.1016/j.ijcard.2011.01.019. Epub 2011 Feb 3. No abstract available. PMID 21295362
- [Background] Te ALD, Wu TC, Lin YJ, Chen YY, Chung FP, Chang SL, Lo LW, Hu YF, Tuan TC, Chao TF, Liao JN, Chien KL, Lin CY, Chang YT, Chen SA. Increased risk of ventricular tachycardia and cardiovascular death in patients with myocarditis during the long-term follow-up: A national representative cohort from the National Health Insurance Research Database. Medicine (Baltimore). 2017 May;96(18):e6633. doi: 10.1097/MD.0000000000006633. PMID 28471960
- [Background] Kang M, An J. Viral Myocarditis. [Updated 2019 Mar 8]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK459259
- [Background] Wojnicz R, Nowalany-Kozielska E, Wojciechowska C, Glanowska G, Wilczewski P, Niklewski T, Zembala M, Polonski L, Rozek MM, Wodniecki J. Randomized, placebo-controlled study for immunosuppressive treatment of inflammatory dilated cardiomyopathy: two-year follow-up results. Circulation. 2001 Jul 3;104(1):39-45. doi: 10.1161/01.cir.104.1.39. PMID 11435335
- [Background] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965
- [Background] From AM, Maleszewski JJ, Rihal CS. Current status of endomyocardial biopsy. Mayo Clin Proc. 2011 Nov;86(11):1095-102. doi: 10.4065/mcp.2011.0296. PMID 22033254
- [Background] Dweck MR, Abgral R, Trivieri MG, Robson PM, Karakatsanis N, Mani V, Palmisano A, Miller MA, Lala A, Chang HL, Sanz J, Contreras J, Narula J, Fuster V, Padilla M, Fayad ZA, Kovacic JC. Hybrid Magnetic Resonance Imaging and Positron Emission Tomography With Fluorodeoxyglucose to Diagnose Active Cardiac Sarcoidosis. JACC Cardiovasc Imaging. 2018 Jan;11(1):94-107. doi: 10.1016/j.jcmg.2017.02.021. Epub 2017 Jun 14. PMID 28624396
- [Background] Wicks EC, Menezes LJ, Barnes A, Mohiddin SA, Sekhri N, Porter JC, Booth HL, Garrett E, Patel RS, Pavlou M, Groves AM, Elliott PM. Diagnostic accuracy and prognostic value of simultaneous hybrid 18F-fluorodeoxyglucose positron emission tomography/magnetic resonance imaging in cardiac sarcoidosis. Eur Heart J Cardiovasc Imaging. 2018 Jul 1;19(7):757-767. doi: 10.1093/ehjci/jex340. PMID 29319785
- [Background] Kadkhodayan A, Chareonthaitawee P, Raman SV, Cooper LT. Imaging of Inflammation in Unexplained Cardiomyopathy. JACC Cardiovasc Imaging. 2016 May;9(5):603-17. doi: 10.1016/j.jcmg.2016.01.010. PMID 27151523
- [Background] Merken J, Hazebroek M, Van Paassen P, Verdonschot J, Van Empel V, Knackstedt C, Abdul Hamid M, Seiler M, Kolb J, Hoermann P, Ensinger C, Brunner-La Rocca HP, Poelzl G, Heymans S. Immunosuppressive Therapy Improves Both Short- and Long-Term Prognosis in Patients With Virus-Negative Nonfulminant Inflammatory Cardiomyopathy. Circ Heart Fail. 2018 Feb;11(2):e004228. doi: 10.1161/CIRCHEARTFAILURE.117.004228. PMID 29449368
- [Background] Frustaci A, Chimenti C. Immunosuppressive therapy in virus-negative inflammatory cardiomyopathy. Herz. 2012 Dec;37(8):854-8. doi: 10.1007/s00059-012-3694-x. PMID 23080270
- [Background] Chan AK, Dohrmann ML. Management of premature ventricular complexes. Mo Med. 2010 Jan-Feb;107(1):39-43. PMID 20222294
- [Background] Kindermann I, Barth C, Mahfoud F, Ukena C, Lenski M, Yilmaz A, Klingel K, Kandolf R, Sechtem U, Cooper LT, Bohm M. Update on myocarditis. J Am Coll Cardiol. 2012 Feb 28;59(9):779-92. doi: 10.1016/j.jacc.2011.09.074. PMID 22361396
- [Background] Fabre A, Sheppard MN. Sudden adult death syndrome and other non-ischaemic causes of sudden cardiac death. Heart. 2006 Mar;92(3):316-20. doi: 10.1136/hrt.2004.045518. Epub 2005 May 27. PMID 15923280
- [Background] Vial T, Descotes J. Immunosuppressive drugs and cancer. Toxicology. 2003 Apr 1;185(3):229-40. doi: 10.1016/s0300-483x(02)00612-1. PMID 12581698
- [Background] Singh JA, Hossain A, Kotb A, Wells G. Risk of serious infections with immunosuppressive drugs and glucocorticoids for lupus nephritis: a systematic review and network meta-analysis. BMC Med. 2016 Sep 13;14(1):137. doi: 10.1186/s12916-016-0673-8. PMID 27623861
- [Background] Kaushik A, Jaimini A, Tripathi M, D'Souza M, Sharma R, Mondal A, Mishra AK, Dwarakanath BS. Estimation of radiation dose to patients from (18) FDG whole body PET/CT investigations using dynamic PET scan protocol. Indian J Med Res. 2015 Dec;142(6):721-31. doi: 10.4103/0971-5916.174563. PMID 26831421
- [Background] Hill MA. Cardiac MR imaging genotoxicity? Eur Heart J. 2018 Jan 21;39(4):313-315. doi: 10.1093/eurheartj/ehx719. No abstract available. PMID 29281062
- [Background] Podrid PJ. Safety and toxicity of antiarrhythmic drug therapy: benefit versus risk. J Cardiovasc Pharmacol. 1991;17 Suppl 6:S65-73. PMID 1723122